CLINICAL TRIAL: NCT05986253
Title: BioDulse II: The Effect of an Irish Seaweed Protein Extract on Glucose Control in Adults With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 23_05_07_EHS
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: A two arm, acute, randomised, double blind, placebo controlled, crossover design feeding study will be used to establish the impact of co-ingestion of BioDulse (a protein hydrolysate from Irish seaweed) with maltodextrin on postprandial blood glucose and insulin concentrations.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): 0.6g/kg body mass maltodextrin in solution
  Interventions: Dietary Supplement: Maltodextrin
- Protein (Experimental): 0.6g/kg body mass maltodextrin PLUS 0.15g/kg body mass protein from Biodulse, in solution
  Interventions: Dietary Supplement: Seaweed protein; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Seaweed protein — Novel protein extracted from seaweed
  Arms: Protein
Dietary Supplement: Maltodextrin — maltodextrin solution

SUMMARY:
Co-ingesting protein with carbohydrate is an effective way to improve postprandial glucose handling. The investigators have isolated and identified a bioactive protein extracted from seaweed. The investigators aim to explore how varying doses of seaweed protein influence postprandial glycaemia and insulinaemia in a population with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-67

Exclusion Criteria:

* Terminal disease
* Exclusively receiving enteral or parenteral nutrition
* Any conditions/anomalies that are contraindications to bioelectrical impedance analysis as per institutional risk assessment and standard operating procedures
* Past medical history of cancer, neurological, kidney, pulmonary, digestive (Coeliac disease), thyroidal disease, cognitive impairment

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Postprandial blood glucose area under the curve (AUC) | 120 minutes
  Integrated area under curve of blood glucose concentration (measured as mmol/L) over 120 minutes

SECONDARY OUTCOMES:
Timecourse of blood glucose concentration | 0, 15, 30, 45, 60, 90, 120 minutes
  Timecourse of blood glucose concentration (measured as mmol/L)
Postprandial serum insulin area under the curve (AUC) | 120 minutes
  Integrated area under curve of blood glucose concentration (measured as mU/L) over 120 minutes
Postprandial serum insulin concentration | 0, 15, 30, 45, 60, 90, 120 minutes
  Timecourse of serum insulin concentration (measured as mU/L)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Carson, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared with researchers outside of those named on the institutional ethics application form.